CLINICAL TRIAL: NCT03733990
Title: A Phase I/II Open-Label, Three-Part, Dose-Finding and Separate Cohort Expansion Trial to Assess the Safety, Tolerability and Preliminary Efficacy of Repeated Doses of CLEVER-1 Antibody FP-1305, in Subjects With Advanced Solid Tumours
Brief Title: A Study to Evaluate Safety, Tolerability and Preliminary Efficacy of FP-1305 in Cancer Patients (MATINS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Faron Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FP2CLI001; 2018-002732-24 (EudraCT Number)
Record Dates: First submitted 2018-10-23; First posted 2018-11-07 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — bexmarilimab

STUDY DESIGN:
Intervention Model Description: Dose-escalation, six dose levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- FP-1305 (bexmarilimab) 0.3 mg/kg (Experimental): Part I, Dose-escalation FP-1305 0.3 mg/kg is administered in Q3W intervals
  Interventions: Biological: FP-1305 (bexmarilimab)
- FP-1305 (bexmarilimab) 1 mg/kg (Experimental): Part I and II, Dose-escalation FP-1305 1 mg/kg is administered in Q3W, Q2W or Q1W intervals
  Interventions: Biological: FP-1305 (bexmarilimab)
- FP-1305 (bexmarilimab) 3 mg/kg (Experimental): Part I and II, Dose-escalation FP-1305 3 mg/kg is administered in Q3W, Q2W or Q1W intervals
  Interventions: Biological: FP-1305 (bexmarilimab)
- FP-1305 (bexmarilimab) 10 mg/kg (Experimental): Part I and II, Dose-escalation FP-1305 10 mg/kg is administered in Q3W, Q2W or Q1W intervals
  Interventions: Biological: FP-1305 (bexmarilimab)
- FP-1305 (bexmarilimab) 0.1 mg/kg (Experimental): Part I Dose-escalation FP-1305 0.1 mg/kg is administered in three-week intervals
  Interventions: Biological: FP-1305 (bexmarilimab)
- FP-1305 (bexmarilimab) 30 mg/kg (Experimental): Part II Dose-escalation FP-1305 30 mg/kg is administered in Q3W, Q2W or Q1W intervals
  Interventions: Biological: FP-1305 (bexmarilimab)

INTERVENTIONS:
Biological: FP-1305 (bexmarilimab) — The study will test for the first time in patients with cancer, an experimental medicine, called FP-1305. The study goal is to find the dose of FP-1305 that works best against cancer while it remains safe for use, tolerable and effective in patients with cancer.
  Other Names: bexmarilimab

SUMMARY:
This is a first in human study to identify whether FP-1305 is suitable to use in humans. The previous pre-clinical studies have demonstrated that FP-1305 binds to a receptor known as CLEVER-1. CLEVER-1 has been shown to support tumour growth. No significant adverse events were witnessed in primates and the dose used will be 300 fold lower than the dose provided to primates which showed no toxicity.

The patients with advanced melanoma, uveal melanoma, cholangiocarcinoma, gallbladder cancer, ER+ breast, gastric, ovarian, pancreatic, colorectal, liver or anaplastic thyroid cancer who have exhausted all licenced therapeutic options will die due to their disease. Based on the investigator's existing data CLEVER-1 is expressed in these tumour types. Inhibition of CLEVER-1 with FP-1305 may have an anti-tumour effect in these patients.

ELIGIBILITY:
Subjects must meet all of the following inclusion criteria to be eligible for participation in the clinical trial:

1. Written Informed Consent
2. Aged ≥ 18 years male or female
3. Tumour sample should be collected during screening period. If a recent tumour biopsy obtained within six months before the date of consent is available (or older, as agreed on a case by case basis with the sponsor), that may be used. At the discretion of the sponsor, the tumour sample may be optional for certain subjects in Part III
4. Life expectancy > 12 weeks
5. Histologically confirmed advanced (inoperable or metastatic) malignancies without standard therapeutic options available:

   * Hepatocellular carcinoma
   * Gallbladder cancer or intra- or extrahepatic cholangiocarcinoma
   * Colorectal adenocarcinoma
   * Serous poorly differentiated (Grade 3) ovarian adenocarcinoma or undifferentiated ovarian cancer
   * Pancreatic ductal adenocarcinoma
   * Immunotherapy (IO) refractory cutaneous melanoma (progression either on or after programmed cell death protein-1 (PD-1)/programmed cell death ligand-1 (PD-L1) or cytotoxic T-lymphocyte antigen-4 (CTLA-4) antibody therapy)
   * Uveal melanoma in Parts II and III
   * Gastric adenocarcinoma (including adenocarcinoma of the distal esophagus / GE junction) in Parts II and III
   * ER+ breast cancer in Parts II and III
   * Anaplastic thyroid cancer in Parts II and III
6. ECOG performance status 0 or 1
7. Measurable disease in Parts II and III
8. Adequate bone marrow, liver and kidney function defined as Blood white blood cell ≥ lower limit of normal Blood neutrophil count ≥ 1x10(9)/L Blood platelet count ≥ 100x10(9)/L, for HCC ≥ 50x10(9)/L Blood haemoglobin ≥ 9.0 g/dL Creatinine clearance > 40 mL/min calculated by Cockcroft-Gault formula AST ≤ 3 X ULN (≤ 5 x ULN when HCC or hepatic metastases are present) ALT ≤ 3 X ULN (≤ 5 x ULN when HCC or hepatic metastases present) Bilirubin ≤ 1.5 X ULN Albumin ≥ 3.0 g/dL The most recent measurements taken during the screening period must be within the required limits for the patient to be considered eligible (i.e. criteria met once during the screening period are not sufficient if there are more recent measurements available that are not within the required limits. It is however acceptable to repeat measurements if the initial measurements or subsequent measurements taken during the screening period are not within the required limits; the patient is eligible providing that the newest measurements are within the required limits). However, once a subject is out of the screening period, and has had eligibility confirmed and been enrolled, the pre-dose laboratory assessments are not subjected to inclusion criteria limits, but only for investigators assessment of subject safety.
9. Women of child-bearing potential must have a negative pregnancy test in serum prior to trial entry
10. Women of child-bearing potential and men who have partners of child-bearing potential must be willing to practise highly effective contraception for the duration of the trial and for three months after the completion of treatment

Exclusion Criteria;

1. Less than 21 days since the last dose of intravenous anticancer chemotherapy or less than five half-lives from a small molecule targeted therapy or oral anticancer chemotherapy before the first IMP administration
2. Any immunotherapy within preceding 6 weeks from the first IMP administration
3. Investigational therapy or major surgery within 4 weeks from the date of consent
4. Active clinically serious infection > Grade 2 NCI-CTCAE version 5.0 (Appendix 5 - Common Toxicity Criteria Gradings) within preceding 2 weeks from the date of consent
5. Brain metastases
6. Subject has not recovered from the previous therapies to Grade ≤ 1 severity as classified by the NCI-CTCAE version 5.0 (except Grade ≤ 2 alopecia, neuropathy or thyroid disorders)
7. Pregnant or lactating women
8. History of second malignancy except for non-melanotic skin cancer, cervical carcinoma in situ or superficial bladder cancer, or any other malignancy treated previously with curative intent and more than three years without relapse
9. Evidence of severe or uncontrolled systemic diseases, congestive cardiac failure New York Heart Association (NYHA) class 2 (Appendix 7 - NYHA classification), Myocardial Infarction (MI) within 6 months or laboratory finding that in the view of the investigator makes it undesirable for the subject to participate in the trial
10. Any medical condition that the Investigator considers significant to compromise the safety of the subject or that impairs the interpretation of IMP toxicity assessment
11. Confirmed human immunodeficiency virus infection
12. Symptomatic cytomegalovirus infection
13. Subjects with active auto-immune disorder (except type I diabetes, celiac disease, hypothyroidism requiring only hormone replacement, vitiligo, psoriasis, or alopecia)
14. The subject requires systemic corticosteroid or other immunosuppressive treatment
15. Subjects with organ transplants
16. Subjects in dialysis
17. Use of Live (attenuated) vaccines for 30 days prior to the start of study treatment, during treatment, and until last visit
18. Subject is unwilling or unable to comply with treatment and trial instructions
19. Subjects with known hypersensitivity to the IMP or any of the pharmaceutical ingredients

Specific Additional Exclusion Criteria for Hepatobiliary Cancers

1. Any ablative therapy (Radio Frequency Ablation or Percutaneous Ethanol Injection) for HCC (this should not exclude subjects if target lesion(s) have not been treated and occurred > 6 weeks prior trial entry)
2. Hepatic encephalopathy
3. Ascites refractory to diuretic therapy
4. Child-Pugh score ≥ 7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petri Bono, MD, PhD, Principal Investigator — Terveystalo Ltd
Locations (11):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States
- Finland (4):
  - Clinical Research Institute HUCH Ltd, Helsinki
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- The Institut Gustave Roussy, Villejuif, France
- Erasmus University Medical Center Rotterdam, Rotterdam, Netherlands
- START Madrid - CIOCC Hospital HM Sanchinarro, Madrid, Spain
- United Kingdom (3):
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rannikko JH, Verlingue L, de Miguel M, Pasanen A, Robbrecht D, Skytta T, Iivanainen S, Shetty S, Ma YT, Graham DM, Arora SP, Jaakkola P, Yap C, Xiang Y, Mandelin J, Karvonen MK, Jalkanen J, Karaman S, Koivunen JP, Minchom A, Hollmen M, Bono P. Bexmarilimab-induced macrophage activation leads to treatment benefit in solid tumors: The phase I/II first-in-human MATINS trial. Cell Rep Med. 2023 Dec 19;4(12):101307. doi: 10.1016/j.xcrm.2023.101307. Epub 2023 Dec 5. PMID 38056464
- [Derived] Hollmen M, Maksimow M, Rannikko JH, Karvonen MK, Vainio M, Jalkanen S, Jalkanen M, Mandelin J. Nonclinical Characterization of Bexmarilimab, a Clever-1-Targeting Antibody for Supporting Immune Defense Against Cancers. Mol Cancer Ther. 2022 Jul 5;21(7):1207-1218. doi: 10.1158/1535-7163.MCT-21-0840. PMID 35500016
- [Derived] Virtakoivu R, Rannikko JH, Viitala M, Vaura F, Takeda A, Lonnberg T, Koivunen J, Jaakkola P, Pasanen A, Shetty S, de Jonge MJA, Robbrecht D, Ma YT, Skytta T, Minchom A, Jalkanen S, Karvonen MK, Mandelin J, Bono P, Hollmen M. Systemic Blockade of Clever-1 Elicits Lymphocyte Activation Alongside Checkpoint Molecule Downregulation in Patients with Solid Tumors: Results from a Phase I/II Clinical Trial. Clin Cancer Res. 2021 Aug 1;27(15):4205-4220. doi: 10.1158/1078-0432.CCR-20-4862. Epub 2021 Jun 2. PMID 34078651

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FP-1305 (Bexmarilimab) 0.3 mg/kg | FP-1305 (Bexmarilimab) 1 mg/kg | FP-1305 (Bexmarilimab) 3 mg/kg | FP-1305 (Bexmarilimab) 10 mg/kg | FP-1305 (Bexmarilimab) 0.1 mg/kg | FP-1305 (Bexmarilimab) 30 mg/kg
Started | 13 | 130 | 41 | 18 | 5 | 9
Completed | 13 | 130 | 41 | 18 | 5 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FP-1305 (Bexmarilimab) 0.3 mg/kg | FP-1305 (Bexmarilimab) 1 mg/kg | FP-1305 (Bexmarilimab) 3 mg/kg | FP-1305 (Bexmarilimab) 10 mg/kg | FP-1305 (Bexmarilimab) 0.1 mg/kg | FP-1305 (Bexmarilimab) 30 mg/kg | Total
Number analyzed (Participants) | 13 | 130 | 41 | 18 | 5 | 9 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 91 | 25 | 9 | 3 | 8 | 139
  >=65 years | 10 | 39 | 16 | 9 | 2 | 1 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.15 (5.444) | 59.67 (10.563) | 61.80 (11.023) | 61.44 (13.321) | 57.60 (16.950) | 57.33 (6.690) | 60.53 (10.787)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 60 | 19 | 6 | 5 | 6 | 104
  Male | 5 | 70 | 22 | 12 | 0 | 3 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race collected as per Sponsor requirements
  Participants
    Asian | 1 | 1 | 0 | 1 | 0 | 0 | 3
    White | 10 | 106 | 33 | 12 | 5 | 8 | 174
    Not reported | 0 | 5 | 1 | 0 | 0 | 0 | 6
    Other | 2 | 18 | 7 | 5 | 0 | 1 | 33
Region of Enrollment [Number; unit: participants]
  Netherlands | 2 | 16 | 8 | 4 | 0 | 1 | 31
  United States | 0 | 4 | 0 | 1 | 0 | 0 | 5
  Finland | 6 | 43 | 12 | 3 | 5 | 3 | 72
  United Kingdom | 5 | 21 | 8 | 3 | 0 | 0 | 37
  France | 0 | 26 | 5 | 4 | 0 | 0 | 35
  Spain | 0 | 20 | 8 | 3 | 0 | 5 | 36

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLT) in the Trial Subjects.
Description: Tolerable dose(s) will be determined by the TITE-CRM based on the occurrence/non-occurrence of dose limiting toxicities in the trial subjects.
Time Frame: Up to one year
Measure: Number; unit: DLT
Arm/Group | FP-1305 (Bexmarilimab) 0.3 mg/kg | FP-1305 (Bexmarilimab) 1 mg/kg | FP-1305 (Bexmarilimab) 3 mg/kg | FP-1305 (Bexmarilimab) 10 mg/kg | FP-1305 (Bexmarilimab) 0.1 mg/kg | FP-1305 (Bexmarilimab) 30 mg/kg
Number analyzed (Participants) | 13 | 130 | 41 | 18 | 5 | 9
DLT | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (Safety and Tolerability)
Description: Number of adverse events and serious adverse events. Adverse events are collected, graded and reported according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Time Frame: approximately 4 years and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1305 (Bexmarilimab) 0.3 mg/kg | FP-1305 (Bexmarilimab) 1 mg/kg | FP-1305 (Bexmarilimab) 3 mg/kg | FP-1305 (Bexmarilimab) 10 mg/kg | FP-1305 (Bexmarilimab) 0.1 mg/kg | FP-1305 (Bexmarilimab) 30 mg/kg
Number analyzed (Participants) | 13 | 130 | 41 | 18 | 5 | 9
Participants | 13 | 122 | 38 | 17 | 5 | 9

3. Primary Outcome: The Response Objective Response Rate (ORR) to the Treatment Was Planned to be Determined by Tumor Imaging According to RECIST 1.1.
Description: The objective response rate (ORR) to the treatment will be determined by tumour imaging (tumor size) according to RECIST v.1.1. Results from each tumour type, dose level and dosing frequency are reported separately.
Time Frame: approximately 4 years and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1305 (Bexmarilimab) 0.3 mg/kg | FP-1305 (Bexmarilimab) 1 mg/kg | FP-1305 (Bexmarilimab) 3 mg/kg | FP-1305 (Bexmarilimab) 10 mg/kg | FP-1305 (Bexmarilimab) 0.1 mg/kg | FP-1305 (Bexmarilimab) 30 mg/kg
Number analyzed (Participants) | 13 | 130 | 41 | 18 | 5 | 9
Participants | 1 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: The Disease Control Rate (DCR) Response to the Treatment Was Planned to be Determined by Tumor Imaging According to RECIST 1.1.
Description: The disease control rate (DCR) response to the treatment will be determined by tumour imaging (tumor size) according to RECIST v.1.1 are presented by cycles and by doing so there is no difference in the definition of DCR and Clinical Benefit Rate (CBR)
Time Frame: approximately 4 years and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | FP-1305 (Bexmarilimab) 0.3 mg/kg | FP-1305 (Bexmarilimab) 1 mg/kg | FP-1305 (Bexmarilimab) 3 mg/kg | FP-1305 (Bexmarilimab) 10 mg/kg | FP-1305 (Bexmarilimab) 0.1 mg/kg | FP-1305 (Bexmarilimab) 30 mg/kg
Number analyzed (Participants) | 13 | 130 | 41 | 18 | 5 | 9
Participants | 1 | 20 | 4 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Approximately 4 years and 11 months
Description: As per clinicaltrials.gov's adverse event definition
Arm/Group | FP-1305 (Bexmarilimab) 0.3 mg/kg | FP-1305 (Bexmarilimab) 1 mg/kg | FP-1305 (Bexmarilimab) 3 mg/kg | FP-1305 (Bexmarilimab) 10 mg/kg | FP-1305 (Bexmarilimab) 0.1 mg/kg | FP-1305 (Bexmarilimab) 30 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/13 | 12/130 | 3/41 | 3/18 | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/13 | 57/130 | 13/41 | 10/18 | 3/5 | 4/9
Other Adverse Events (participants affected / at risk) | 13/13 | 122/130 | 38/41 | 17/18 | 5/5 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FP-1305 (Bexmarilimab) 0.3 mg/kg (N=13) | FP-1305 (Bexmarilimab) 1 mg/kg (N=130) | FP-1305 (Bexmarilimab) 3 mg/kg (N=41) | FP-1305 (Bexmarilimab) 10 mg/kg (N=18) | FP-1305 (Bexmarilimab) 0.1 mg/kg (N=5) | FP-1305 (Bexmarilimab) 30 mg/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Ascites (Gastrointestinal disorders) | 0 | 5 (7) | 2 (2) | 1 (1) | 2 (2) | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 5 (5) | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 (3) | 2 (2) | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 (2) | 0 | 0 | 0 | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 1 (2) | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (2) | 1 (1) | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 3 (3) | 3 (3) | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 (3) | 1 (1) | 0 | 1 (1) | 0
General physical health deterioration (General disorders) | 0 | 2 (2) | 0 | 0 | 1 (1) | 0
Fatigue (General disorders) | 0 | 1 (2) | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 (1) | 0 | 2 (2) | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 (2) | 1 (1) | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Infected seroma (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Infection (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 3 (3) | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 (2) | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 (2) | 0 | 1 (1) | 0 | 0
Abdominal pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 | 0 | 0 | 0
Metastases to oesophagus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1) | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1) | 0 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 1 (2) | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 (4) | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FP-1305 (Bexmarilimab) 0.3 mg/kg (N=13) | FP-1305 (Bexmarilimab) 1 mg/kg (N=130) | FP-1305 (Bexmarilimab) 3 mg/kg (N=41) | FP-1305 (Bexmarilimab) 10 mg/kg (N=18) | FP-1305 (Bexmarilimab) 0.1 mg/kg (N=5) | FP-1305 (Bexmarilimab) 30 mg/kg (N=9)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (3) | 32 (52) | 11 (15) | 6 (11) | 1 (1) | 2 (2)
Cardiac disorders (Cardiac disorders) | 0 | 3 (7) | 1 (1) | 1 (1) | 0 | 0
Endocrine disorders (Endocrine disorders) | 1 (3) | 4 (4) | 0 | 0 | 0 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 7 (13) | 49 (145) | 20 (44) | 5 (22) | 2 (11) | 5 (8)
General disorders and administration site conditions (General disorders) | 8 (15) | 57 (99) | 16 (24) | 11 (16) | 3 (6) | 6 (8)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2) | 7 (16) | 3 (4) | 1 (1) | 0 | 0
Infections and infestations (Infections and infestations) | 2 (3) | 16 (22) | 7 (11) | 1 (2) | 2 (3) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 5 (8) | 3 (4) | 1 (1) | 0 | 1 (1)
Investigations (Investigations) | 4 (10) | 40 (104) | 10 (22) | 6 (18) | 2 (7) | 3 (7)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (5) | 36 (55) | 10 (26) | 8 (12) | 1 (1) | 0
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 (10) | 25 (47) | 12 (18) | 5 (8) | 1 (2) | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 9 (11) | 4 (5) | 2 (3) | 1 (1) | 0
Nervous system disorders (Nervous system disorders) | 3 (5) | 14 (25) | 6 (14) | 1 (1) | 0 | 6 (6)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 7 (8) | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 21 (30) | 4 (5) | 3 (3) | 1 (1) | 1 (3)
Vascular disorders (Vascular disorders) | 0 | 13 (13) | 5 (5) | 2 (5) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03733990/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT03733990/SAP_001.pdf